CLINICAL TRIAL: NCT00540501
Title: Phase 1, Open-Label Study to Evaluate Potential Pharmacokinetic Interactions Between Orally-Administered Oseltamivir and Intravenous Zanamivir in Healthy Thai Adult Subjects
Brief Title: A Study to Evaluate Orally-Administered Oseltamivir and Intravenous Zanamivir in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Contract agreement not reached
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAI108166
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Subjects
Keywords: zanamivir,; influenza virus,; healthy volunteer,; PK, drug interaction,; IV, and oseltamivir.
MeSH Terms: interventions — Oseltamivir

ARMS (4):
- Oseltamivir 150mg and zanamivir 50mg/hour (Experimental): Oseltamivir1 150mg PO q12h for 5 doses + Zanamivir IV continuous infusion at 50mg/hour for 72 hours
  Interventions: Drug: Oseltamivir and Intravenous Zanamivir
- Zanamivir IV 50mg/hour (Experimental): Zanamivir IV continuous infusion 50mg/hour for 16 hours (total dose of 800mg)
  Interventions: Drug: Oseltamivir and Intravenous Zanamivir
- Oseltamivir 150mg and zanamivir 600mg (Experimental): Oseltamivir 150mg PO q12h for 5 doses + Zanamivir 600mg IV q12h
  Interventions: Drug: Oseltamivir and Intravenous Zanamivir
- Oseltamivir 150mg (Active Comparator): Oseltamivir 150mg PO q12h for 3 days
  Interventions: Drug: Oseltamivir and Intravenous Zanamivir

INTERVENTIONS:
Drug: Oseltamivir and Intravenous Zanamivir — Oseltamivir will be administered PO q12h for 3 days (for a total of 5 doses ending the morning of day 3.
  Both drugs will be administered simultaneously starting on Day 1 of Period 3. Zanamivir will be administered IV q12h for 3 days (for a total of 5 doses ending on the morning of day 3.
  Zanamivir to be given four (4) hours after the oral dose of oseltamivir and infused over 30 minutes.

SUMMARY:
This study is a 4 period study to see if there is any interaction between Orally-Administered Oseltamivir and Intravenous Zanamivir in Healthy Thai Adult Subjects

ELIGIBILITY:
Inclusion criteria:

* Healthy Volunteer(s)confirmed by physical exam, clinical labs, ECGs, and vitals
* Must be woman of non-childbearing potential or willing to abstain from intercourse for two weeks prior to study drug administration and throughout the study or be willing to use two acceptable methods of birth control.

Exclusion criteria:

* Subjects with history of certain heart problems or subjects with Hepatitis B, C or HIV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Estimated); Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Oseltamivir carboxylate levels: Cmax and AUC(0-12)- | Period 2: Day 1, 2 & 3. Period 3: Day 1, 2 & 3. Period 4: Day 1, 2 & 3.

SECONDARY OUTCOMES:
Oseltamivir: Cmax, AUC(0-12)& C12. Oseltamivir carboxylate: C12, AUC(0-24)& t1/2. | Period 2-4 Day 1-3
Zanamivir: Cmax, AUC(0-12), C12, t1/2, CL, tmax & V2 . | Period 1, 3 & 4 Day 1-3
Safety:labs, vitals, ECGs & AEs. | Period 1-4, Days 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline